CLINICAL TRIAL: NCT02700477
Title: Clinical Evaluation of Fenugreek Seed Extract In Patients With Type- 2 Diabetes: An Add-On Study
Brief Title: Evaluation of Fenugreek Seed Extract In Type- 2 Diabetes: An Add-On Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chemical Resources (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: Protocol No. CR001/02/13
Record Dates: First submitted 2015-09-29; First posted 2016-03-07 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-03

CONDITIONS: Diabetes
Keywords: Type-2 Diabetic; HbA1c; FBS; PPBS; C-peptide
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fenugreek seed extract (Active Comparator): Fenugreek seeds extract 500 mg capsule twice a day for 12 weeks
  Interventions: Dietary Supplement: Fenugreek seeds extract
- Placebo (Placebo Comparator): Placebo capsule containing Dicalcium Phosphate 500mg, BD
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Fenugreek seeds extract — Fenugreek seed extract 500mg, BD
  Other Names: Fenfuro
  Arms: Fenugreek seed extract
Other: Placebo — Placebo capsule containing Dicalcium Phosphate 500mg, BD
  Arms: Placebo

SUMMARY:
Trigonella Foenum-Graecum, commonly known as Fenugreek, is a plant that has been extensively used as a source of anti-diabetic compounds Fenugreek is traditionally used in India, especially in the Ayurvedic and Unani systems.

Preliminary animal and human trials suggest possible hypoglycemic and anti-hyper lipidemic properties of Fenugreek seed powder, when taken orally. Fenugreek seeds contain 50% fiber (30% soluble fiber and 20% insoluble fiber) that can slow the rate of post-prandial glucose absorption. This may be a secondary mechanism for the hypoglycemic effect.

DETAILED DESCRIPTION:
Diabetes mellitus is a complex heterogeneous group of metabolic conditions characterized by increased levels of blood glucose due to impairment in insulin action and/or insulin secretion. Diabetes is a condition primarily defined by the level of hyperglycemia giving rise to risk of microvascular damage (retinopathy, nephropathy and neuropathy). It is associated with reduced life expectancy, significant morbidity due to specific diabetes related Microvascular complications, increased risk of macrovascular complications (ischemic heart disease, stroke and peripheral vascular disease), and diminished quality of life.Type 2 diabetes mellitus (T2DM) is the most common form of diabetes in humans and results from a combination of genetic and acquired factors that impair -cell function and tissue insulin sensitivity.

The WHO has put the number of persons with diabetes worldwide at approximately 170 million. The prevalence of diabetes mellitus has risen dramatically over the past 20 years, and the number of people with diabetes is expected to reach 366 million by 2025. The prevalence of type 2 diabetes mellitus is expected to grow even more rapidly in the future. There is also considerable geographic variation in the incidence of T2DM, and countries like India are fast emerging as ''diabetes hot spots". About 5-10% of the total health care budget has been used for T2DM in many countries.

Reduced pancreatic β-cell functional mass in diabetes, and other categories of glucose intolerance, has been described by several authors, and decreased islet and/or -cell volume in the pancreas of type 2 diabetic patients has been consistently reported. In addition, studies conducted in patients, and isolated islets, have shown both quantitative and qualitative defects of glucose-stimulated insulin secretion.

The ideal antidiabetic agent should normalize plasma glucose, minimize side effects, and prevent development of micro- and macrovascular complications. Obviously no such agent is available, nor is it likely to be available in the near or medium-term future.

Current treatments and treatment regimens include combinations of oral antidiabetic drugs (OADs), antihypertensive medications, and antidyslipidemic agents, but these have been less than successful in managing their respective disease targets with clinical goals. Measures such as screening and intensive life-style modification can help to delay the onset of diabetes in at-risk individuals, and stringent glycemic control with pharmacotherapy may improve outcomes. To manage the type 2 diabetes epidemic effectively, however, agents that can effectively and durably controls glycemia while providing pleiotropic benefits (e.g. blood pressure reduction) are required.

The landmark Diabetes Control and Complications Trial and the United Kingdom Prospective Diabetes Study (UKPDS) have convincingly demonstrated that normalizing glycosylated hemoglobin (HbA1C) levels in individuals with diabetes can reduce diabetes-related cardio-vascular (CV) morbidity and mortality as well as the incidence and progression of micro vascular complications.

HbA1C concentration is an accurate predictor of risk for such complications, with a desirable goal of 7.0% or less. In the clinical setting, measurement of HbA1C assesses longer-term glycemic control among individuals with diabetes.

A range of therapeutic agents exist for the treatment of type 2 diabetes. Metformin, a biguanide, is a commonly prescribed oral anti diabetic drug; American Diabetes Association (ADA)/European Association for the Study of Diabetes (EASD) guidelines recommend metformin as initial pharmacotherapy for type 2 diabetes, with an expected reduction in HbA1C of between 1.0% and 2.0%. In their recommendations, both the ADA and the International Diabetes Foundation support metformin as initial pharmacotherapy for type 2 diabetes.

However, Metformin is associated with increased CV risk and lactic acidosis, and it is contraindicated in patients with heart failure or impaired renal function. Metformin monotherapy has also been associated with diarrhea in approximately 50% of patients and nausea or vomiting in 25% of patients.

Sulfonylurea's (SUs) e.g., glimepiride have long been an effective and low-cost mainstay of type 2 diabetes therapy; as with metformin, SU monotherapy can be expected to reduce HbA1C by 1.0% to 2.0%. SUs are a common alternative or add-on to metformin and act by stimulating pancreatic beta-cell insulin secretion in a glucose-independent manner. Weight gain is a common adverse effect of SU therapy, as is an increased risk of hypoglycemia, particularly in the elderly and in patients with worsening renal function.

Thiazolidinedione (TZD) monotherapy has been associated with HbA1C reductions of between 0.5% and 1.4%. TZDs have beneficial effects on CV markers, including lipid levels (particularly triglycerides and HDL-Cholesterol), blood pressure, inflammatory mediators, endothelial function, and fibrinolytic status. However, weight gain and increased risk of edema and heart failure are frequent adverse effects, particularly when TZDs are used in combination with insulin.

Alpha-glucosidase inhibitors, such as acarbose, act as competitive inhibitors of the alpha glucosidases, thereby delaying glucose absorption. This effect on glucose uptake decreases glucose peak and insulin response postprandially and moderately lowers fasting plasma glucose levels and HbA1C, but gastrointestinal adverse effects and the requirement for three times daily dosing may inhibit adherence to therapy. Monotherapy with alpha-glucosidase inhibitors have been associated with HbA1C reductions of between 0.5% and 0.8%, with no weight gain.

Glinide (i.e., repaglinide, nateglinide) monotherapy has been reported to reduce HbA1C by between 0.5% and 1.5%. The rapid onset of action of glinides necessitates three times daily dosing, and they have been associated with hypoglycemia. Weight gain has been reported with glinide therapy (between 0.7 and 1.8 kg).

Insulin, either alone or in combination with other agents, most commonly metformin, is an effective option for restoring normoglycemia, especially when administered early in the disease course. The disadvantages of insulin therapy are weight gain and an increased risk of hypoglycemia. Insulin has not been observed to have clinically relevant effects on either blood pressure or lipids.

In addition to devising the most appropriate pharmacotherapeutic regimen for the patient with type 2 diabetes, patient management is also of critical importance and is best handled by a medical care team including the physician, the pharmacist, the dietitian, and a diabetes education specialist. Ideally, a diabetes care plan should be developed with input from all medical care team practitioners and the patient. Incretin-based therapies, which include the glucagon-like peptide (GLP)-1 receptor agonist's exenatide and exenatide Long acting release (LAR), and liraglutide and the Dipeptidyl peptidase-4 (DPP-4) inhibitors sitagliptin, vildagliptin, and saxagliptin represent a new class of antidiabetic drugs. Data suggest an equal or potentially greater efficacy of incretin-based therapies to lower HbA1C compared with other antidiabetic therapies, with a low risk of hypoglycemia. Other benefits include weight reduction (GLP-1 receptor agonists) or weight neutrality (DPP-4 inhibitors).GLP-1 receptor agonists have recently been added to the ADA/EASD treatment algorithm as a tier 2 alternative to the addition of SUs or basal insulin in patients not adequately controlled on metformin plus lifestyle modification.

The OADs are able, for a time, to reduce A1C but do not correct all the metabolic and glucoregulatory dysfunctions involved in type 2 diabetes pathophysiology. As a result, HbA1C goals become more difficult to maintain and a significant glycemic burden accumulates, increasing the risk of CV diseases. The treatment of co morbid conditions, particularly hypertension, may also impede achieving and maintaining glycemic goals. Difficulties in maintaining long-term glycemic control with currently available antidiabetic therapies have led to the need for additional treatments that can be used as monotherapy or combined safely with existing agents and that may target more of the underlying pathologies of type 2 diabetes.

Although traditional treatments and treatment combinations are initially successful at lowering HbA1C, they are unable to restore normoglycemia over the long term. Recent data that suggest the mean time to secondary failure on OADs (a therapeutic event necessitating the addition of another agent or insulin) may be as short as 1.3 years.

The primary goal in the treatment of patients with type 2 diabetes is the maintenance of beta-cell function, the decline of which is the major reason for impairment in glucose tolerance over time. Consequently, therapies that arrest progressive beta-cell deterioration while restoring and maintaining normoglycemia will be required. New therapies are needed that will also minimize weight gain and correct dyslipidemia without compromising improvements in glycemic control.

The Investigational Agent Trigonella Foenum Graecum, commonly known as Fenugreek, is a plant that has been extensively used as a source of antidiabetic compounds, from its seeds, leaves and extracts in different model systems. Fenugreek is traditionally used in India, especially in the Ayurvedic and Unani systems.Preliminary animal and human trials suggest possible hypoglycemic and anti-hyperlipidemic properties of fenugreek seed powder taken orally. Fenugreek seeds contain 50% fiber (30% soluble fiber and 20% insoluble fiber) that can slow the rate of post-prandial glucose absorption. This may be a secondary mechanism for the hypoglycemic effect.

ELIGIBILITY:
Inclusion Criteria:

* Either gender & Attending diabetic clinical at hospital
* Type-2 DM <5 years duration
* On oral hypoglycaemic agents( Metformin±Sulfonylurea)
* No change in anti-diabetic treatment for the last one month
* HbA1c >7.5%
* Fasting plasma glucose not exceeding 180mg/dL
* Patient able to make proper use of medication.
* Patients willing to provide signed informed consent

Exclusion Criteria:

* Diabetes other than type 2 diabetes mellitus
* Evidence of renal disease (Serum creatinine > 1.5mg/ml)
* Evidence of liver disease (aspartate transaminase (AST) and alanine transaminase (ALT) >3 times of normal)
* Pregnant and lactating mothers and women intending pregnancy
* Participation in any other clinical trial with in the last 30 days
* History of any hemoglobinopathy that may affect determination of Glycosylated Haemoglobin
* Treatment with oral anti-diabetic agents (other than Metformin or SU) during the 12 weeks before baseline visit.
* History of intolerance or hypersensitivity to sulfonylurea or Metformin or Fenugreek seed extract.
* Any condition which in the opinion of the PI is significant and can make the patient unsuitable for study or can place it under additional risk.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 154 (Actual)
Dates: Start 2013-07; Primary Completion 2014-05 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Fasting blood sugar levels | 12 weeks
  Reduction in fasting blood sugar levels (FBS) (mg/dL)
Post prandial blood sugar levels | 12 weeks
  Reduction in post prandial blood sugar levels (mg/dL)

SECONDARY OUTCOMES:
Glycosylated haemoglobin (HbA1C)(%) | 12 weeks
  Reduction in glycosylated haemoglobin

CONTACTS AND LOCATIONS:
Overall Officials: Dr Narsingh Verma, MD, Principal Investigator — Dept of Physiology,King George's Medical University, Lucknow, UP, India

REFERENCES:
- [Background] Chehade JM, Gladysz M, Mooradian AD. Dyslipidemia in type 2 diabetes: prevalence, pathophysiology, and management. Drugs. 2013 Mar;73(4):327-39. doi: 10.1007/s40265-013-0023-5. PMID 23479408
- [Result] Verma R, Khanna P, Mehta B. National programme on prevention and control of diabetes in India: Need to focus. Australas Med J. 2012;5(6):310-5. doi: 10.4066/AMJ.2012.1340. Epub 2012 Jun 30. No abstract available. PMID 22848329